CLINICAL TRIAL: NCT01584843
Title: A Multicenter, Randomized, Evaluator-masked, Parallel-group, Non-treatment-controlled Study Followed by an Open-label Study to Evaluate Efficacy and Safety of GSK1358820 (Botulinum Toxin Type A) in Patients With Strabismus
Brief Title: Efficacy and Safety of GSK1358820 (Botulinum Toxin Type A) in Patients With Strabismus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 116246
Record Dates: First submitted 2012-04-23; First posted 2012-04-25 (Estimated); Results first posted 2014-08-01 (Estimated); Last update posted 2015-07-24 (Estimated); Status verified 2015-03

CONDITIONS: Strabismus
Keywords: Neuromuscular Agents; Strabismus; Botulinum Toxin Type A
MeSH Terms: conditions — Strabismus | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Non-treatment (10-20 PD) (No Intervention): Receive no treatment on Week 0
- GSK1358820 1.25 U (10-20 PD) (Active Comparator): Receive 1.25 U of GSK1358820 on Week 0
  Interventions: Drug: GSK1358820
- GSK1358820 2.5 U (10-20 PD) (Active Comparator): Receive 2.5 U of GSK1358820 on Week 0
  Interventions: Drug: GSK1358820
- Non-treatment (20-50 PD) (No Intervention): Receive no treatment on Week 0
- GSK1358820 2.5 U (20-50 PD) (Active Comparator): Receive 2.5 U of GSK1358820 on Week 0
  Interventions: Drug: GSK1358820
- GSK1358820 5.0 U (20-50 PD) (Active Comparator): Receive 5.0 U of GSK1358820 on Week 0
  Interventions: Drug: GSK1358820

INTERVENTIONS:
Drug: GSK1358820 — IM injection of Botulinum Toxin Type A
  Other Names: Botulinum Toxin Type A
  Arms: GSK1358820 1.25 U (10-20 PD); GSK1358820 2.5 U (10-20 PD); GSK1358820 2.5 U (20-50 PD); GSK1358820 5.0 U (20-50 PD)

SUMMARY:
Primary objective is to evaluate the efficacy of single-dose treatment with GSK1358820 compared with non-treatment in patients with strabismus based on angles of strabismus in the primary position.

DETAILED DESCRIPTION:
Primary objective is to evaluate the efficacy of single-dose treatment with GSK1358820 compared with non-treatment in patients with strabismus based on angles of strabismus in the primary position. Secondary objective is to evaluate the efficacy and safety of repeated-dose treatment with GSK1358820 in patients with strabismus.

ELIGIBILITY:
Inclusion Criteria:

<At the start of screening period>

* Paralytic or concomitant strabismus. Subjects with paralytic strabismus will be eligible for inclusion only if paralysis has persisted for at least 3 months and strabismus has been developed at one eye
* Horizontal deviations (esotropia or exotropia)
* Strabismus with the (absolute) strabismus angles at both distance and near of primary position >-10 PD and <50 PD
* Age>-12 years at the time of giving informed consent
* The subject has to be capable of giving written informed consent of their own will. For subjects aged less than 20 years, the subject and his/her legally acceptable representative (person in parental authority or guardian) have to give written informed consent
* Either sex. Males have to agree to practice contraception during the study period. Females of child-bearing potential will be eligible for inclusion in this study. However, they have to have negative pregnancy test both at the screening visit and just before initial injection and agree to practice reliable methods of contraception
* QTc <450 msec; for patients with Bundle Branch Block, QTc <480 msec based on average QTc value of triplicate ECGs <At the start of treatment period >
* Strabismus with the (absolute) strabismus angles at both distance and near of primary position >-10 PD and <50 PD
* ALT at the screening visit <2 x ULN and alkaline phosphatase and bilirubin <-1.5 x ULN

Exclusion Criteria:

<At the start of screening period>

* Secondary strabismus caused by prior surgical recession of the antagonist in past surgical treatment of strabismus
* Strabismus due to abnormal innervations
* Strabismus with thyroid-associated ophthalmopathy
* Strabismus with strong motor limitation of extraocular muscles
* Mechanical limitations of ocular movement due to periorbital disease or due to past surgical treatment other than strabismus
* Blepharoptosis
* Conjunctival pathology
* Systemic neuromuscular junction dysfunction
* Systemic neuromuscular disease
* Past treatment with botulinum toxin
* Planned injections of botulinum toxin for other indication(s) or for cosmetic purpose during the study period
* Known hypersensitivity to any of the drugs to be used in the study or history of allergy
* Treatment with antibiotics with neuromuscular junction inhibitory action such as aminoglycosides, polypeptides, tetracyclines and lincomycins, except those contained in topical antibacterial formulations
* Treatment with muscle relaxants or drugs with muscle relaxant action
* Chronic respiratory disorder
* Severe muscle weakness or atrophy
* Angle-closure glaucoma or its predisposing factors
* Severe cardiac, hepatic or renal impairment. The severity refers to Grade 3 according to "the Classification of the Severity of Adverse Experiences" (MHLW PAB/SD Notification No. 80, dated 29 June 1992).
* Surgical operation or hospitalization to be needed during the study period
* Female subjects who are pregnant or lactating, who may be pregnant, or who plan for pregnancy during the study period
* Participation in another clinical study within 6 months prior to enrollment in this study or planned participation in another clinical study after enrollment in this study
* Psychiatric disorder or impairment of intellectual function that may affect the subject's ability to give informed consent or to comply with the trial procedures
* History of alcohol dependence or drug abuse
* Subjects whom the investigator (or sub-investigator) considers ineligible for the study

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2012-05; Primary Completion 2013-07 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (10):
- Japan (10):
  - GSK Investigational Site, Aichi
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Hyōgo
  - GSK Investigational Site, Kagoshima
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Miyazaki
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Shizuoka
  - GSK Investigational Site, Tokyo
  - GSK Investigational Site, Yamaguchi

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study consisted of a Screening Period (1-2 weeks), the First Treatment Period (12-52 weeks), and the Second Treatment Period (24 weeks). In this summary, data are presented for participants who completed Week 24 of the First Treatment Period.
Pre-assignment Details: A total of 41 participants with horizontal strabismus meeting the selection criteria were divided into two strata in terms of the mean of the distant-view strabismus angle and the near-view strabismus angle in the primary position: >=10 prism dioptre (PD) to <20 PD as Strata 1 and >=20 PD to <50 PD as Strata 2.
Groups:
- BSA >=10 PD and <20 PD: Non-treatment, Then GSK1358820: Participants (Par) with a Baseline strabismus angle (BSA) >=10 prism dioptre (PD) and <20 PD received no treatment at the start of the First Treatment Period (FTP). Par who met the additional injection criteria at 4 weeks after the start of the FTP received the injection of GSK1358820, either 1.25 Units (U) or 2.5 U, at one site of the medial rectus muscle or the lateral rectus muscle of the affected eye, then were observed for 12-24 weeks. Par who met the re-injection criteria at 12-24 weeks after the last injection (of the FTP) entered the Second Treatment Period (STP) to receive the re-injection at an appropriate dose level selected by the investigator from the prior dose level, then were observed for 24 weeks. Par who did not meet the re-injection criteria were observed for 24 more weeks. Par received a maximum of 2 injections.
- BSA >=10 PD and <20 PD: GSK1358820 1.25 U: Par with a BSA >=10 PD and <20 PD received the first injection of GSK1358820 1.25 U at one site of the medial rectus muscle or the lateral rectus muscle of the affected eye at the start of the FTP. Par who met the additional injection criteria at 4 weeks after the start of the FTP received an additional injection of GSK1358820, either 1.25 U or 2.5 U, at the same site and in the same eye as the previous injection, then were observed for 12-24 weeks. Par who met the re-injection criteria at 12-24 weeks after the last injection (of the FTP) entered the STP to receive the re-injection at an appropriate dose level selected by the investigator from the prior dose level, then were observed for 24 weeks. Par who did not meet the re-injection criteria were observed for 24 more weeks. Par received a maximum of 3 injections.
- BSA >=10 PD and <20 PD: GSK1358820 2.5 U: Par with a BSA >=10 PD and <20 PD received the first injection of GSK1358820 2.5 U at one site of the medial rectus muscle or the lateral rectus muscle of the affected eye at the start of the FTP. Par who met the additional injection criteria at 4 weeks after the start of the FTP received an additional injection of GSK1358820, either 2.5 U or 5.0 U, at the same site and in the same eye as the previous injection, then were observed for 12-24 weeks. Par who met the re-injection criteria at 12-24 weeks after the last injection (of the FTP) entered the STP to receive the re-injection at an appropriate dose level selected by the investigator from the prior dose level, then were observed for 24 weeks. Par who did not meet the re-injection criteria were observed for 24 more weeks. Par received a maximum of 3 injections.
- BSA >=20 PD and <50 PD: Non-treatment, Then GSK1358820: Par with a BSA >=20 PD and <50 PD received no treatment at the start of the FTP. Par who met the additional injection criteria at 4 weeks after the start of the FTP received the injection of GSK1358820, either 2.5 U or 5.0 U, at one site of the medial rectus muscle or the lateral rectus muscle of the affected eye, then were observed for 12-24 weeks. Par who met the re-injection criteria at 12-24 weeks after the last injection (of the FTP) entered the STP to receive the re-injection at an appropriate dose level selected by the investigator from the prior dose level, then were observed for 24 weeks. Par who did not meet the re-injection criteria were observed for 24 more weeks. Par received a maximum of 2 injections.
- BSA >=20 PD and <50 PD: GSK1358820 2.5 U: Par with a BSA >=20 PD and <50 PD received the first injection of GSK1358820 2.5 U at one site of the medial rectus muscle or the lateral rectus muscle of the affected eye at the start of the FTP. Par who met the additional injection criteria at 4 weeks after the start of the FTP received an additional injection of GSK1358820, either 2.5 U or 5.0, at the same site and in the same eye as the previous injection, then were observed for 12-24 weeks. Par who met the re-injection criteria at 12-24 weeks after the last injection (of the FTP) entered the STP to receive the re-injection at an appropriate dose level selected by the investigator from the prior dose level, then were observed for 24 weeks. Par who did not meet the re-injection criteria were observed for 24 more weeks. Par received a maximum of 3 injections.
- BSA >=20 PD and <50 PD: GSK1358820 5.0 U: Par with a BSA >=20 PD and <50 PD received the first injection of GSK1358820 5.0 U at one site of the medial rectus muscle or the lateral rectus muscle of the affected eye at the start of the FTP. Par who met the additional injection criteria at 4 weeks after the start of the FTP received an additional injection of GSK1358820, either 5.0 U or 10.0 U, at the same site and in the same eye as the previous injection, then were observed for 12-24 weeks. Par who met the re-injection criteria at 12-24 weeks after the last injection (of the FTP) entered the STP to receive the re-injection at an appropriate dose level selected by the investigator from the prior dose level, then were observed for 24 weeks. Par who did not meet the re-injection criteria were observed for 24 more weeks. Par received a maximum of 3 injections.
Period: First Treatment Period
Arm/Group | BSA >=10 PD and <20 PD: Non-treatment, Then GSK1358820 | BSA >=10 PD and <20 PD: GSK1358820 1.25 U | BSA >=10 PD and <20 PD: GSK1358820 2.5 U | BSA >=20 PD and <50 PD: Non-treatment, Then GSK1358820 | BSA >=20 PD and <50 PD: GSK1358820 2.5 U | BSA >=20 PD and <50 PD: GSK1358820 5.0 U
Started | 3 | 4 | 3 | 10 | 10 | 11
Completed | 3 | 4 | 2 | 10 | 10 | 9
Not Completed | 0 | 0 | 1 | 0 | 0 | 2
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Met Protocol-defined Stopping Criteria | 0 | 0 | 0 | 0 | 0 | 1
Period: Second Treatment Period
Arm/Group | BSA >=10 PD and <20 PD: Non-treatment, Then GSK1358820 | BSA >=10 PD and <20 PD: GSK1358820 1.25 U | BSA >=10 PD and <20 PD: GSK1358820 2.5 U | BSA >=20 PD and <50 PD: Non-treatment, Then GSK1358820 | BSA >=20 PD and <50 PD: GSK1358820 2.5 U | BSA >=20 PD and <50 PD: GSK1358820 5.0 U
Started | 2 | 1 | 2 | 6 | 3 | 1
Completed | 2 | 1 | 2 | 6 | 3 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Non-treatment, Then GSK1358820: Participants (par) with a Baseline strabismus angle (BSA) >=10 prism dioptre (PD) and <20 PD or with a BSA >=20 PD and <50 PD received no treatment from the start of the First Treatment Period (FTP). Par who met the additional injection criteria at 4 weeks after the start of the FTP received the injection of GSK1358820, either 1.25 Units (U), 2.5 U, or 5.0 U at one site of the medial rectus muscle or the lateral rectus muscle of the affected eye, then were observed for 12-24 weeks. Par who met the re-injection criteria at 12-24 weeks after the last injection (of the FTP) entered the Second Treatment Period (STP) to receive the re-injection at an appropriate dose level selected by the investigator from the prior dose level, then were observed for 24 weeks. Par who did not meet the re-injection criteria were observed for 24 more weeks. Par received a maximum of 2 injections.
- GSK1358820 1.25 U: Par with a BSA >=10 PD and <20 PD received the first injection of GSK1358820 1.25 U at one site of the medial rectus muscle or the lateral rectus muscle of the affected eye at the start of the FTP. Par who met the additional injection criteria at 4 weeks after the start of the FTP received an additional injection of GSK1358820, either 1.25 U or 2.5 U, at the same site and in the same eye as the previous injection, then were observed for 12-24 weeks. Par who met the re-injection criteria at 12-24 weeks after the last injection (of the FTP) entered the STP to receive the re-injection at an appropriate dose level selected by the investigator from the prior dose level, then were observed for 24 weeks. Par who did not meet the re-injection criteria were observed for 24 more weeks. Par received a maximum of 3 injections.
- GSK1358820 2.5 U: Par with a BSA >=10 PD and <20 PD or with a BSA >=20 PD and <50 PD received the first injection of GSK1358820 2.5 U at one site of the medial rectus muscle or the lateral rectus muscle of the affected eye at the start of the FTP. Par who met the additional injection criteria at 4 weeks after the start of the FTP received an additional injection of GSK1358820, either 2.5 U or 5.0 U, at the same site and in the same eye as the previous injection, then were observed for 12-24 weeks. Par who met the re-injection criteria at 12-24 weeks after the last injection (of the FTP) entered the STP to receive the re-injection at an appropriate dose level selected by the investigator from the prior dose level, then were observed for 24 weeks. Par who did not meet the re-injection criteria were observed for 24 more weeks. Par received a maximum of 3 injections.
- GSK1358820 5.0 U: Par with a BSA >=20 PD and <50 PD received the first injection of GSK1358820 5.0 U at one site of the medial rectus muscle or the lateral rectus muscle of the affected eye at the start of the FTP. Par who met the additional injection criteria at 4 weeks after the start of the FTP received an additional injection of GSK1358820, either 5.0 U or 10.0 U, at the same site and in the same eye as the previous injection, then were observed for 12-24 weeks. Par who met the re-injection criteria at 12-24 weeks after the last injection (of the FTP) entered the STP to receive the re-injection at an appropriate dose level selected by the investigator from the prior dose level, then were observed for 24 weeks. Par who did not meet the re-injection criteria were observed for 24 more weeks. Par received a maximum of 3 injections.
- Total: Total of all reporting groups
Arm/Group | Non-treatment, Then GSK1358820 | GSK1358820 1.25 U | GSK1358820 2.5 U | GSK1358820 5.0 U | Total
Number analyzed (Participants) | 13 | 4 | 13 | 11 | 41
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.5 (23.67) | 19.8 (9.07) | 51.4 (22.78) | 49.0 (21.79) | 45.1 (23.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 3 | 7 | 5 | 22
  Male | 6 | 1 | 6 | 6 | 19
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian - Japanese Heritage | 13 | 4 | 13 | 11 | 41

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Strabismus Angle Prism Dioptre (PD) in the Primary Position at Week 4 of the FTP in Observed Cases (OC)
Description: The strabismus angle in the primary position was measured using the alternative prism cover test (APCT). The strabismus angle was evaluated as the mean value of the distant-view strabismus angle (measured at a distance of 5 meters [m]) and the near-view strabismus angle (measured at a distance of 33 centimeters [cm]). Every participant's evaluation was performed in the same affected eye (left or right) throughout the study period. Change from Baseline was calculated as the value at Week 4 minus the value at Baseline.
Time Frame: Baseline and Week 4 of the FTP
Population: Full Analysis Set (FAS1) Population: all participants who were randomized and had at least one post-Baseline efficacy assessment. Values were summarized for OC of the FTP without imputation of missing values. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: prism dioptre
Groups:
- SA >=20 PD and <50 PD: Non-treatment, Then GSK1358820: Par with a BSA >=20 PD and <50 PD received no treatment at the start of the FTP. Par who met the additional injection criteria at 4 weeks after the start of the FTP received the injection of GSK1358820, either 2.5 U or 5.0 U, at one site of the medial rectus muscle or the lateral rectus muscle of the affected eye, then were observed for 12-24 weeks. Par who met the re-injection criteria at 12-24 weeks after the last injection (of the FTP) entered the STP to receive the re-injection at an appropriate dose level selected by the investigator from the prior dose level, then were observed for 24 weeks. Par who did not meet the re-injection criteria were observed for 24 more weeks. Par received a maximum of 2 injections.
Arm/Group | BSA >=10 PD and <20 PD: Non-treatment, Then GSK1358820 | BSA >=10 PD and <20 PD: GSK1358820 1.25 U | BSA >=10 PD and <20 PD: GSK1358820 2.5 U | SA >=20 PD and <50 PD: Non-treatment, Then GSK1358820 | BSA >=20 PD and <50 PD: GSK1358820 2.5 U | BSA >=20 PD and <50 PD: GSK1358820 5.0 U
Number analyzed (Participants) | 3 | 4 | 2 | 10 | 10 | 11
prism dioptre | 2.33 (6.602) | -7.50 (7.141) | -3.75 (2.475) | -0.55 (2.291) | -13.40 (15.105) | -17.27 (15.476)
Statistical Analysis 1: Comparison: BSA >=10 PD and <20 PD: Non-treatment, Then GSK1358820 vs BSA >=10 PD and <20 PD: GSK1358820 1.25 U; Test type: Superiority or Other; p = 0.091, Fisher LSD method — LSD=Least Significant Difference; Mean Difference (Final Values) = -9.83, 95% CI 2-sided [-21.81 to 2.14]
Statistical Analysis 2: Comparison: BSA >=10 PD and <20 PD: Non-treatment, Then GSK1358820 vs BSA >=10 PD and <20 PD: GSK1358820 2.5 U; Test type: Superiority or Other; p = 0.338, Fisher LSD method; Mean Difference (Final Values) = -6.08, 95% CI 2-sided [-20.39 to 8.23]
Statistical Analysis 3: Comparison: BSA >=10 PD and <20 PD: GSK1358820 1.25 U vs BSA >=10 PD and <20 PD: GSK1358820 2.5 U; Test type: Superiority or Other; p = 0.524, Fisher LSD method; Mean Difference (Final Values) = 3.75, 95% CI 2-sided [-9.83 to 17.33]
Statistical Analysis 4: Comparison: SA >=20 PD and <50 PD: Non-treatment, Then GSK1358820 vs BSA >=20 PD and <50 PD: GSK1358820 2.5 U; Test type: Superiority or Other; p = 0.031, Fisher LSD method; Mean Difference (Final Values) = -12.85, 95% CI 2-sided [-24.46 to -1.24]
Statistical Analysis 5: Comparison: SA >=20 PD and <50 PD: Non-treatment, Then GSK1358820 vs BSA >=20 PD and <50 PD: GSK1358820 5.0 U; Test type: Superiority or Other; p = 0.005, Fisher LSD method; Mean Difference (Final Values) = -16.72, 95% CI 2-sided [-28.06 to -5.38]
Statistical Analysis 6: Comparison: BSA >=20 PD and <50 PD: GSK1358820 2.5 U vs BSA >=20 PD and <50 PD: GSK1358820 5.0 U; Test type: Superiority or Other; p = 0.490, Fisher LSD method; Mean Difference (Final Values) = -3.87, 95% CI 2-sided [-15.21 to 7.47]

2. Secondary Outcome: Change From Baseline in the Strabismus Angle Prism Dioptre (PD) in the Primary Position at Week 1 After the Initial Injection of the FTP in Observed Cases (OC)
Description: The strabismus angle in the primary position was measured using the APCT. The strabismus angle was evaluated as the mean value of the distant-view strabismus angle (measured at a distance of 5 m) and the near-view strabismus angle (measured at a distance of 33 cm). Every participant's evaluation was performed in the same affected eye (left or right) throughout the study period. Change from Baseline was calculated as the value at Week 1minus the value at Baseline.
Time Frame: Baseline and Week 1 of the FTP
Population: FAS1 Population
Measure: Mean (Standard Deviation); unit: prism dioptre
Arm/Group | BSA >=10 PD and <20 PD: Non-treatment, Then GSK1358820 | BSA >=10 PD and <20 PD: GSK1358820 1.25 U | BSA >=10 PD and <20 PD: GSK1358820 2.5 U | BSA >=20 PD and <50 PD: Non-treatment, Then GSK1358820 | BSA >=20 PD and <50 PD: GSK1358820 2.5 U | BSA >=20 PD and <50 PD: GSK1358820 5.0 U
Number analyzed (Participants) | 3 | 4 | 3 | 10 | 10 | 11
prism dioptre | 1.50 (1.323) | -5.75 (8.180) | 8.83 (19.902) | -1.70 (3.285) | -16.35 (20.033) | -19.73 (11.376)

3. Secondary Outcome: Change From Baseline in the Strabismus Angle PD in the Primary Position at Weeks 1, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, and 48 After the Final Injection of the FTP
Description: The strabismus angle in the primary position was measured using the APCT. The strabismus angle was evaluated as the mean value of the distant-view strabismus angle (measured at a distance of 5 m) and the near-view strabismus angle (measured at a distance of 33 cm). Every participant's evaluation was performed in the same affected eye (left or right) throughout the study period. The values were summarized for the observed cases for the change in the strabismus angle in the primary position from Baseline at Weeks 1, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44 and 48 (before reinjection of the second treatment period if applicable) after the final injection of the FTP (after randomization in the non-treatment groups). Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline and Weeks 1, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, and 48 after the final injection of the FTP
Population: FAS1 Population
Measure: Mean (Standard Deviation); unit: prism dioptre
Arm/Group | BSA >=10 PD and <20 PD: Non-treatment, Then GSK1358820 | BSA >=10 PD and <20 PD: GSK1358820 1.25 U | BSA >=10 PD and <20 PD: GSK1358820 2.5 U | BSA >=20 PD and <50 PD: Non-treatment, Then GSK1358820 | BSA >=20 PD and <50 PD: GSK1358820 2.5 U | BSA >=20 PD and <50 PD: GSK1358820 5.0 U
Number analyzed (Participants) | 3 | 4 | 3 | 10 | 10 | 11
prism dioptre
  Week 1, n=3, 4, 3, 10, 10, 11 | -8.17 (2.566) | -5.75 (8.180) | 5.83 (22.115) | -11.15 (8.307) | -16.35 (20.033) | -22.36 (14.063)
  Week 4, n=3, 4, 2, 10, 10, 11 | -6.83 (3.329) | -7.50 (7.141) | -3.75 (8.132) | -11.90 (5.092) | -13.15 (15.324) | -19.55 (16.378)
  Week 8, n=3, 4, 2, 10, 10, 10 | -4.50 (2.291) | -7.50 (6.245) | 2.00 (2.828) | -8.90 (5.934) | -8.85 (10.588) | -13.50 (16.074)
  Week 12, n=3, 4, 2, 10, 10, 10 | -2.83 (6.788) | -5.00 (7.439) | 2.50 (9.899) | -7.65 (4.090) | -6.00 (6.811) | -12.95 (13.150)
  Week 16, n=2, 4, 2, 9, 10, 10 | -5.75 (1.768) | -4.88 (10.103) | -1.75 (3.889) | -6.50 (5.990) | -7.65 (8.573) | -11.60 (16.244)
  Week 20, n=2, 4, 0, 7, 9, 9 | -5.75 (1.768) | -4.63 (8.845) | NA (NA) — No participants in this treatment arm were analyzed at this time point. | -6.21 (4.091) | -6.00 (6.933) | -10.28 (11.514)
  Week 24, n=1, 3, 0, 5, 8, 9 | -5.00 (NA) — The standard deviation cannot be calculated because only one participant was analyzed in this treatment arm at this time point. | -7.33 (11.579) | NA (NA) — No participants in this treatment arm were analyzed at this time point. | -3.40 (2.679) | -8.31 (8.422) | -10.28 (12.171)
  Week 28, n=1, 3, 0, 4, 7, 8 | -4.00 (NA) — The standard deviation cannot be calculated because only one participant was analyzed in this treatment arm at this time point. | -5.17 (11.751) | NA (NA) — No participants in this treatment arm were analyzed at this time point. | -5.63 (4.191) | -6.86 (9.335) | -10.31 (16.722)
  Week 32, n=1, 3, 0, 4, 7, 8 | -2.00 (NA) — The standard deviation cannot be calculated because only one participant was analyzed in this treatment arm at this time point. | -4.67 (13.650) | NA (NA) — No participants in this treatment arm were analyzed at this time point. | -2.38 (2.056) | -6.29 (8.401) | -9.94 (12.486)
  Week 36, n=1, 3, 0, 4, 7, 8 | -2.00 (NA) — The standard deviation cannot be calculated because only one participant was analyzed in this treatment arm at this time point. | -3.33 (13.503) | NA (NA) — No participants in this treatment arm were analyzed at this time point. | -4.75 (4.213) | -5.50 (9.363) | -8.38 (15.784)
  Week 40, n=1, 3, 0, 4, 7, 8 | -4.00 (NA) — The standard deviation cannot be calculated because only one participant was analyzed in this treatment arm at this time point. | -2.83 (12.332) | NA (NA) — No participants in this treatment arm were analyzed at this time point. | -1.50 (3.629) | -7.00 (11.206) | -10.19 (14.909)
  Week 44, n=1, 3, 0, 4, 7, 8 | -4.00 (NA) — The standard deviation cannot be calculated because only one participant was analyzed in this treatment arm at this time point. | -1.00 (14.000) | NA (NA) — No participants in this treatment arm were analyzed at this time point. | -2.00 (7.382) | -6.79 (9.725) | -9.25 (14.378)
  Week 48, n=1, 3, 0, 4, 7, 8 | -2.00 (NA) — The standard deviation cannot be calculated because only one participant was analyzed in this treatment arm at this time point. | -1.33 (13.796) | NA (NA) — No participants in this treatment arm were analyzed at this time point. | -1.00 (4.546) | -9.21 (7.521) | -9.94 (10.722)

4. Secondary Outcome: Change From Baseline in the Strabismus Angle PD in the Primary Position at Weeks 1, 4, 8, 12, 16, 20, and 24 of the Second Treatment Period (STP)
Description: The strabismus angle in the primary position was measured using the APCT. The strabismus angle was evaluated as the mean value of the distant-view strabismus angle (measured at a distance of 5 m) and the near-view strabismus angle (measured at a distance of 33 cm). Every participant's evaluation was performed in the same affected eye (left or right) throughout the study period. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline and Weeks 1, 4, 8, 12, 16, 20, and 24 of the STP (up to Study Week 52)
Population: FAS2 Population: all participants who were included in the FAS1 Population, received reinjection of the investigational product, and had at least one efficacy assessment after the reinjection
Measure: Mean (Standard Deviation); unit: prism dioptre
Arm/Group | BSA >=10 PD and <20 PD: Non-treatment, Then GSK1358820 | BSA >=10 PD and <20 PD: GSK1358820 1.25 U | BSA >=10 PD and <20 PD: GSK1358820 2.5 U | BSA >=20 PD and <50 PD: Non-treatment, Then GSK1358820 | BSA >=20 PD and <50 PD: GSK1358820 2.5 U | BSA >=20 PD and <50 PD: GSK1358820 5.0 U
Number analyzed (Participants) | 2 | 1 | 2 | 6 | 3 | 1
prism dioptre
  Week 1, n=2, 1, 2, 6, 3, 1 | -2.75 (12.374) | -1.00 (NA) — The standard deviation cannot be calculated because there were not enough participants analyzed in this treatment arm at this time point | -7.75 (1.061) | -16.08 (9.641) | -7.83 (7.006) | -9.50 (NA) — The standard deviation cannot be calculated because there were not enough participants analyzed in this treatment arm at this time point
  Week 4, n=2, 1, 2, 6, 3, 1 | -5.25 (7.425) | -3.00 (NA) — The standard deviation cannot be calculated because there were not enough participants analyzed in this treatment arm at this time point | -6.75 (5.303) | -11.25 (9.010) | -11.83 (1.756) | -6.50 (NA) — The standard deviation cannot be calculated because there were not enough participants analyzed in this treatment arm at this time point
  Week 8, n=2, 1, 2, 6, 3, 0 | -0.75 (10.960) | -3.00 (NA) — The standard deviation cannot be calculated because there were not enough participants analyzed in this treatment arm at this time point | 2.75 (11.667) | -12.33 (13.717) | -10.00 (3.122) | NA (NA) — No participants in this treatment arm were analyzed at this time point
  Week 12, n=2, 1, 2, 6, 3, 1 | -1.25 (10.253) | 1.00 (NA) — The standard deviation cannot be calculated because there were not enough participants analyzed in this treatment arm at this time point | 1.25 (3.889) | -10.17 (7.421) | -7.67 (2.517) | -4.50 (NA) — The standard deviation cannot be calculated because there were not enough participants analyzed in this treatment arm at this time point
  Week 16, n=1, 1, 2, 6, 3, 0 | 6.00 (NA) — The standard deviation cannot be calculated because there were not enough participants analyzed in this treatment arm at this time point | -2.00 (NA) — The standard deviation cannot be calculated because there were not enough participants analyzed in this treatment arm at this time point | 3.25 (4.596) | -6.75 (8.413) | -5.83 (3.819) | NA (NA) — No participants in this treatment arm were analyzed at this time point
  Week 20, n=2, 1, 2, 6, 3, 0 | -1.25 (10.253) | -2.00 (NA) — The standard deviation cannot be calculated because there were not enough participants analyzed in this treatment arm at this time point | 0.50 (7.071) | -7.42 (9.308) | -2.00 (6.083) | NA (NA) — No participants in this treatment arm were analyzed at this time point
  Week 24, n=1, 1, 2, 6, 3, 0 | 2.50 (NA) — The standard deviation cannot be calculated because there were not enough participants analyzed in this treatment arm at this time point | -2.00 (NA) — The standard deviation cannot be calculated because there were not enough participants analyzed in this treatment arm at this time point | 0.50 (0.707) | -6.83 (7.387) | -2.33 (4.752) | NA (NA) — No participants in this treatment arm were analyzed at this time point

5. Secondary Outcome: Absolute Strabismus Angle in the Primary Position at Weeks 1 and 4 of the FTP
Description: The strabismus angle in the primary position was measured using the APCT. The strabismus angle was evaluated as the mean value of the distant-view strabismus angle (measured at a distance of 5 m) and the near-view strabismus angle (measured at a distance of 33 cm). Every participant's evaluation was performed in the same affected eye (left or right) throughout the study period. The absolute values of the strabismus angle in the primary position at Week 1 and Week 4 of the FTP were summarized for observed cases without imputation of missing values.
Time Frame: Weeks 1 and 4 of the FTP
Population: FAS1 Population
Measure: Mean (Standard Deviation); unit: prism dioptre
Arm/Group | BSA >=10 PD and <20 PD: Non-treatment, Then GSK1358820 | BSA >=10 PD and <20 PD: GSK1358820 1.25 U | BSA >=10 PD and <20 PD: GSK1358820 2.5 U | BSA >=20 PD and <50 PD: Non-treatment, Then GSK1358820 | BSA >=20 PD and <50 PD: GSK1358820 2.5 U | BSA >=20 PD and <50 PD: GSK1358820 5.0 U
Number analyzed (Participants) | 3 | 4 | 3 | 10 | 10 | 11
prism dioptre
  Week 1, n=3, 4, 3, 10, 10, 11 | 17.67 (2.754) | 9.25 (7.182) | 24.00 (18.358) | 32.05 (9.385) | 14.20 (21.953) | 15.55 (16.090)
  Week 4, n=3, 4, 2, 10, 10, 11 | 18.50 (7.794) | 7.50 (6.137) | 12.00 (1.414) | 33.20 (9.855) | 17.15 (17.645) | 18.00 (18.126)

6. Secondary Outcome: Absolute Strabismus Angle in the Primary Position at Weeks 1, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, and 48 After the Final Injection of the FTP
Description: The strabismus angle in the primary position was measured using the APCT. The strabismus angle was evaluated as the mean value of the distant-view strabismus angle (measured at a distance of 5 m) and the near-view strabismus angle (measured at a distance of 33 cm). Every participant's evaluation was performed in the same affected eye (left or right) throughout the study period. The absolute values of the strabismus angle in the primary position were summarized for observed cases at Weeks 1, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, and 48 (before reinjection of the second treatment period if applicable) after the final injection of the FTP (after randomization in the non-treatment groups).
Time Frame: Weeks 1, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, and 48 after the final injection of the FTP
Population: FAS1 Population
Measure: Mean (Standard Deviation); unit: prism dioptre
Arm/Group | BSA >=10 PD and <20 PD: Non-treatment, Then GSK1358820 | BSA >=10 PD and <20 PD: GSK1358820 1.25 U | BSA >=10 PD and <20 PD: GSK1358820 2.5 U | BSA >=20 PD and <50 PD: Non-treatment, Then GSK1358820 | BSA >=20 PD and <50 PD: GSK1358820 2.5 U | BSA >=20 PD and <50 PD: GSK1358820 5.0 U
Number analyzed (Participants) | 3 | 4 | 3 | 10 | 10 | 11
prism dioptre
  Week 1, n=3, 4, 3, 10, 10, 11 | 8.00 (1.732) | 9.25 (7.182) | 21.00 (20.809) | 22.60 (14.261) | 14.20 (21.953) | 12.91 (16.386)
  Week 4, n=3, 4, 2, 10, 10, 11 | 9.33 (4.041) | 7.50 (6.137) | 12.00 (4.243) | 21.85 (11.626) | 17.40 (17.980) | 15.73 (17.934)
  Week 8, n=3, 4, 2, 10, 10, 10 | 11.67 (4.041) | 7.50 (5.323) | 17.75 (1.061) | 24.85 (12.985) | 21.70 (14.442) | 20.95 (18.570)
  Week 12, n=3, 4, 2, 10, 10, 10 | 13.33 (8.737) | 10.00 (6.481) | 18.25 (6.010) | 26.10 (10.501) | 24.55 (10.289) | 21.50 (14.193)
  Week 16, n=2, 4, 2, 9, 10, 10 | 9.50 (4.950) | 10.13 (9.313) | 14.00 (0.000) | 28.50 (12.684) | 22.90 (12.030) | 22.85 (17.626)
  Week 20, n=2, 4, 0, 7, 9, 9 | 9.50 (4.950) | 10.38 (8.138) | NA (NA) — No participants in this treatment arm were analyzed at this time point. | 27.36 (11.775) | 23.50 (9.031) | 23.00 (13.720)
  Week 24, n=1, 3, 0, 5, 8, 9 | 8.00 (NA) — The standard deviation cannot be calculated because only one participant was analyzed in this treatment arm at this time point. | 8.00 (10.966) | NA (NA) — No participants in this treatment arm were analyzed at this time point. | 30.10 (12.577) | 22.38 (9.837) | 23.00 (12.186)
  Week 28, n=1, 3, 0, 4, 7, 8 | 9.00 (NA) — The standard deviation cannot be calculated because only one participant was analyzed in this treatment arm at this time point. | 10.17 (10.797) | NA (NA) — No participants in this treatment arm were analyzed at this time point. | 27.50 (15.199) | 23.57 (11.638) | 24.31 (18.225)
  Week 32, n=1, 3, 0, 4, 7, 8 | 11.00 (NA) — The standard deviation cannot be calculated because only one participant was analyzed in this treatment arm at this time point. | 10.67 (12.897) | NA (NA) — No participants in this treatment arm were analyzed at this time point. | 30.75 (12.639) | 24.14 (10.633) | 24.69 (12.587)
  Week 36, n=1, 3, 0, 4, 7, 8 | 11.00 (NA) — The standard deviation cannot be calculated because only one participant was analyzed in this treatment arm at this time point. | 12.00 (12.530) | NA (NA) — No participants in this treatment arm were analyzed at this time point. | 28.38 (15.617) | 24.93 (12.654) | 26.25 (16.466)
  Week 40, n=1, 3, 0, 4, 7, 8 | 9.00 (NA) — The standard deviation cannot be calculated because only one participant was analyzed in this treatment arm at this time point. | 12.50 (10.966) | NA (NA) — No participants in this treatment arm were analyzed at this time point. | 31.63 (14.739) | 23.43 (14.243) | 24.44 (15.562)
  Week 44, n=1, 3, 0, 4, 7, 8 | 9.00 (NA) — The standard deviation cannot be calculated because only one participant was analyzed in this treatment arm at this time point. | 14.33 (12.662) | NA (NA) — No participants in this treatment arm were analyzed at this time point. | 31.13 (17.731) | 23.64 (12.877) | 25.38 (14.665)
  Week 48, n=1, 3, 0, 4, 7, 8 | 11.00 (NA) — The standard deviation cannot be calculated because only one participant was analyzed in this treatment arm at this time point. | 14.00 (12.490) | NA (NA) — No participants in this treatment arm were analyzed at this time point. | 32.13 (15.644) | 21.21 (9.309) | 24.69 (11.065)

7. Secondary Outcome: Absolute Strabismus Angle in the Primary Position at Weeks 1, 4, 8, 12, 16, 20, and 24 of the STP
Description: The strabismus angle in the primary position was measured using the APCT. The strabismus angle was evaluated as the mean value of the distant-view strabismus angle (measured at a distance of 5 m) and the near-view strabismus angle (measured at a distance of 33 cm). Every participant's evaluation was performed in the same affected eye (left or right) throughout the study period.
Time Frame: Weeks 1, 4, 8, 12, 16, 20, and 24 of the STP (up to Study Week 52)
Population: FAS2 population.
Measure: Mean (Standard Deviation); unit: prism dioptre
Arm/Group | BSA >=10 PD and <20 PD: Non-treatment, Then GSK1358820 | BSA >=10 PD and <20 PD: GSK1358820 1.25 U | BSA >=10 PD and <20 PD: GSK1358820 2.5 U | BSA >=20 PD and <50 PD: Non-treatment, Then GSK1358820 | BSA >=20 PD and <50 PD: GSK1358820 2.5 U | BSA >=20 PD and <50 PD: GSK1358820 5.0 U
Number analyzed (Participants) | 2 | 1 | 2 | 6 | 3 | 1
prism dioptre
  Week 1, n=2, 1, 2, 6, 3, 1 | 15.00 (12.728) | 13.00 (NA) — The standard deviation cannot be calculated because only one participant has been analyzed in this treatment arm at this time point. | 8.00 (2.828) | 18.08 (10.097) | 23.00 (15.395) | 13.00 (NA) — The standard deviation cannot be calculated because only one participant has been analyzed in this treatment arm at this time point.
  Week 4, n=2, 1, 2, 6, 3, 1 | 12.50 (7.778) | 11.00 (NA) — The standard deviation cannot be calculated because only one participant has been analyzed in this treatment arm at this time point. | 9.00 (1.414) | 22.92 (10.646) | 19.00 (11.822) | 16.00 (NA) — The standard deviation cannot be calculated because only one participant has been analyzed in this treatment arm at this time point.
  Week 8, n=2, 1, 2, 6, 3, 0 | 17.00 (11.314) | 11.00 (NA) — The standard deviation cannot be calculated because only one participant has been analyzed in this treatment arm at this time point. | 18.50 (7.778) | 21.83 (12.356) | 20.83 (10.867) | NA (NA) — No participants in this treatment arm were analyzed at this time point.
  Week 12, n=2, 1, 2, 6, 3, 1 | 16.50 (10.607) | 15.00 (NA) — The standard deviation cannot be calculated because only one participant has been analyzed in this treatment arm at this time point. | 17.00 (0.000) | 24.00 (9.690) | 23.17 (11.514) | 18.00 (NA) — The standard deviation cannot be calculated because only one participant has been analyzed in this treatment arm at this time point.
  Week 16, n=1, 1, 2, 6, 3, 0 | 24.00 (NA) — The standard deviation cannot be calculated because only one participant has been analyzed in this treatment arm at this time point. | 12.00 (NA) — The standard deviation cannot be calculated because only one participant has been analyzed in this treatment arm at this time point. | 19.00 (0.707) | 27.42 (11.222) | 25.00 (11.456) | NA (NA) — No participants in this treatment arm were analyzed at this time point.
  Week 20, n=2, 1, 2, 6, 3, 0 | 16.50 (10.607) | 12.00 (NA) — The standard deviation cannot be calculated because only one participant has been analyzed in this treatment arm at this time point. | 16.25 (3.182) | 26.75 (13.171) | 28.83 (15.543) | NA (NA) — No participants in this treatment arm were analyzed at this time point.
  Week 24, n=1, 1, 2, 6, 3, 0 | 20.50 (NA) — The standard deviation cannot be calculated because only one participant has been analyzed in this treatment arm at this time point. | 12.00 (NA) — The standard deviation cannot be calculated because only one participant has been analyzed in this treatment arm at this time point. | 16.25 (4.596) | 27.33 (9.621) | 28.50 (14.807) | NA (NA) — No participants in this treatment arm were analyzed at this time point.

8. Secondary Outcome: Percent Change From Baseline in the Strabismus Angle in the Primary Position at Week 1 and Week 4 in Observed Cases (OC) of the FTP
Description: The strabismus angle in the primary position was measured using the APCT. The strabismus angle was evaluated as the mean value of the distant-view strabismus angle (measured at a distance of 5 m) and the near-view strabismus angle (measured at a distance of 33 cm). Every participant's evaluation was performed in the same affected eye (left or right) throughout the study period. The values were summarized for observed cases for the percent change from Baseline in the strabismus angle in the primary position at Week 1and Week 4 after the initial injection in the FTP. Percent change from Baseline in the strabismus angle was calculated as: absolute angle ([strabismus angle at Baseline minus strabismus angle after the final injection] divided by the absolute strabismus angle at Baseline) multiplied by 100.
Time Frame: Baseline and Weeks 1 and 4 of the FTP
Population: FAS1 Population
Measure: Mean (Standard Deviation); unit: Percent change in prism dioptre
Arm/Group | BSA >=10 PD and <20 PD: Non-treatment, Then GSK1358820 | BSA >=10 PD and <20 PD: GSK1358820 1.25 U | BSA >=10 PD and <20 PD: GSK1358820 2.5 U | BSA >=20 PD and <50 PD: Non-treatment, Then GSK1358820 | BSA >=20 PD and <50 PD: GSK1358820 2.5 U | BSA >=20 PD and <50 PD: GSK1358820 5.0 U
Number analyzed (Participants) | 3 | 4 | 3 | 10 | 10 | 11
Percent change in prism dioptre
  Week 1, n=3, 4, 3, 10, 10, 11 | 9.77 (8.491) [8.491 to -35.98] | -35.98 (48.460) | 68.00 (136.601) | -5.33 (9.956) | -56.91 (67.224) | -61.28 (37.603)
  Week 4, n=3, 4, 2, 10, 10, 11 | 13.50 (36.745) [lower limit 36.745] | -47.98 (42.069) | -22.55 (10.112) | -2.32 (7.337) | -47.19 (51.238) | -52.40 (46.823)

9. Secondary Outcome: Percent Change From Baseline in the Strabismus Angle in the Primary Position at Weeks 1, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, and 48 After the Final Injection of the FTP
Description: The strabismus angle in the primary position was measured using the APCT. The strabismus angle was evaluated as the mean value of the distant-view strabismus angle (measured at a distance of 5 m) and the near-view strabismus angle (measured at a distance of 33 cm). Every participant's evaluation was performed in the same affected eye (left or right) throughout the study period. The values were summarized for observed cases for percent change from Baseline in the strabismus angle in the primary position at Weeks 1, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, and 48 (before reinjection of the second treatment period if applicable) after the final injection of the FTP (after randomization in non-treatment groups; up to a maximum of 52 weeks of the FTP). Percent change from Baseline in the strabismus angle was calculated as: (absolute angle [strabismus angle at Baseline minus the strabismus angle after the final injection] divided by the absolute strabismus angle at Baseline) multiplied by
Time Frame: Baseline and Weeks 1, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, and 48 of the FTP
Population: FAS1 Population
Measure: Mean (Standard Deviation); unit: Percent change in prism dioptre
Arm/Group | BSA >=10 PD and <20 PD: Non-treatment, Then GSK1358820 | BSA >=10 PD and <20 PD: GSK1358820 1.25 U | BSA >=10 PD and <20 PD: GSK1358820 2.5 U | BSA >=20 PD and <50 PD: Non-treatment, Then GSK1358820 | BSA >=20 PD and <50 PD: GSK1358820 2.5 U | BSA >=20 PD and <50 PD: GSK1358820 5.0 U
Number analyzed (Participants) | 3 | 4 | 3 | 10 | 10 | 11
Percent change in prism dioptre
  Week 1, n=3, 4, 3, 10, 10, 11 | -50.07 (9.697) | -35.98 (48.460) | 47.17 (151.828) | -37.64 (27.691) | -56.91 (67.224) | -66.98 (40.186)
  Week 4, n=3, 4, 2, 10, 10, 11 | -42.80 (19.128) | -47.98 (42.069) | -18.00 (47.235) | -38.96 (20.351) | -46.56 (51.832) | -57.80 (46.560)
  Week 8, n=3, 4, 2, 10, 10, 10 | -28.90 (15.431) | -48.43 (35.871) | 15.40 (21.779) | -30.50 (23.971) | -32.40 (34.610) | -41.62 (44.030)
  Week 12, n=3, 4, 2, 10, 10, 10 | -21.03 (43.107) | -31.23 (44.523) | 24.40 (68.872) | -24.69 (14.030) | -21.09 (22.844) | -38.02 (34.387)
  Week 16, n=2, 4, 2, 9, 10, 10 | -39.75 (19.870) | -30.13 (62.986) | -8.30 (22.627) | -22.00 (19.920) | -27.16 (28.721) | -34.80 (39.312)
  Week 20, n=2, 4, 0, 7, 9, 9 | -39.75 (19.870) | -28.93 (55.046) | NA (NA) — No participants in this treatment arm were analyzed at this time point. | -21.60 (17.290) | -20.59 (23.190) | -31.97 (29.371)
  Week 24, n=1, 3, 0, 5, 8, 9 | -38.50 (NA) — The standard deviation cannot be calculated because only one participant was analyzed in this treatment arm at this time point. | -46.10 (72.788) | NA (NA) — No participants in this treatment arm were analyzed at this time point. | -13.32 (13.777) | -27.75 (28.362) | -29.84 (31.502)
  Week 28, n=1, 3, 0, 4, 7, 8 | -30.80 (NA) — The standard deviation cannot be calculated because only one participant was analyzed in this treatment arm at this time point | -30.80 (71.776) | NA (NA) — No participants in this treatment arm were analyzed at this time point. | -21.75 (18.746) | -23.81 (30.638) | -31.00 (41.524)
  Week 32, n=1, 3, 0, 4, 7, 8 | -15.40 (NA) — The standard deviation cannot be calculated because only one participant was analyzed in this treatment arm at this time point | -27.77 (85.545) | NA (NA) — No participants in this treatment arm were analyzed at this time point. | -8.63 (7.602) | -21.53 (27.576) | -28.08 (28.243)
  Week 36, n=1, 3, 0, 4, 7, 8 | -15.40 (NA) — The standard deviation cannot be calculated because only one participant was analyzed in this treatment arm at this time point | -18.23 (83.395) | NA (NA) — No participants in this treatment arm were analyzed at this time point. | -19.65 (20.539) | -20.21 (29.986) | -24.15 (36.602)
  Week 40, n=1, 3, 0, 4, 7, 8 | -30.80 (NA) — The standard deviation cannot be calculated because only one participant was analyzed in this treatment arm at this time point | -13.97 (74.899) | NA (NA) — No participants in this treatment arm were analyzed at this time point. | -8.20 (15.849) | -25.30 (35.381) | -29.48 (33.356)
  Week 44, n=1, 3, 0, 4, 7, 8 | -30.80 (NA) — The standard deviation cannot be calculated because only one participant was analyzed in this treatment arm at this time point | -1.43 (86.222) | NA (NA) — No participants in this treatment arm were analyzed at this time point. | -11.10 (24.612) | -24.39 (30.858) | -26.38 (32.674)
  Week 48, n=1, 3, 0, 4, 7, 8 | -15.40 (NA) — The standard deviation cannot be calculated because only one participant was analyzed in this treatment arm at this time point | -3.80 (84.778) | NA (NA) — No participants in this treatment arm were analyzed at this time point. | -6.78 (14.954) | -30.91 (25.390) | -28.09 (24.167)

10. Secondary Outcome: Percent Change From Baseline in the Strabismus Angle in the Primary Position at Weeks 1, 4, 8, 12, 16, 20, and 24 of the STP
Description: The strabismus angle in the primary position was measured using the APCT. The strabismus angle was evaluated as the mean value of the distant-view strabismus angle (measured at a distance of 5 m) and the near-view strabismus angle (measured at a distance of 33 cm). Every participant's evaluation was performed in the same affected eye (left or right) throughout the study period. Percent change from Baseline in the strabismus angle was calculated as: (absolute angle [strabismus angle at Baseline minus the strabismus angle after the final injection] divided by the absolute strabismus angle at Baseline) multiplied by 100.
Time Frame: Baseline and Weeks 1, 4, 8, 12, 16, 20, and 24 of the STP (up to Study Week 52)
Population: FAS2 Population
Measure: Mean (Standard Deviation); unit: Percent change in prism dioptre
Arm/Group | BSA >=10 PD and <20 PD: Non-treatment, Then GSK1358820 | BSA >=10 PD and <20 PD: GSK1358820 1.25 U | BSA >=10 PD and <20 PD: GSK1358820 2.5 U | BSA >=20 PD and <50 PD: Non-treatment, Then GSK1358820 | BSA >=20 PD and <50 PD: GSK1358820 2.5 U | BSA >=20 PD and <50 PD: GSK1358820 5.0 U
Number analyzed (Participants) | 2 | 1 | 2 | 6 | 3 | 1
Percent change in prism dioptre
  Week 1, n=2, 1, 2, 6, 3, 1 | -16.20 (70.004) | -7.10 (NA) — The standard deviation cannot be calculated because only one participant has been analyzed in this treatment arm at this time point. | -49.85 (5.586) | -46.75 (26.774) | -30.50 (26.754) | -42.20 (NA) — The standard deviation cannot be calculated because only one participant has been analyzed in this treatment arm at this time point.
  Week 4, n=2, 1, 2, 6, 3, 1 | -30.00 (42.426) | -21.40 (NA) — The standard deviation cannot be calculated because only one participant has been analyzed in this treatment arm at this time point. | -39.95 (23.829) | -33.33 (27.466) | -43.13 (21.925) | -28.90 (NA) — The standard deviation cannot be calculated because only one participant has been analyzed in this treatment arm at this time point.
  Week 8, n=2, 1, 2, 6, 3, 0 | -4.85 (61.872) | -21.40 (NA) — The standard deviation cannot be calculated because only one participant has been analyzed in this treatment arm at this time point. | 27.45 (80.822) | -33.95 (32.783) | -35.10 (14.224) | NA (NA) — No participants in this treatment arm were analyzed at this time point.
  Week 12, n=2, 1, 2, 6, 3, 1 | -7.65 (57.912) | 7.10 (NA) — The standard deviation cannot be calculated because only one participant has been analyzed in this treatment arm at this time point. | 11.35 (27.506) | -29.87 (21.927) | -27.77 (13.999) | -20.00 (NA) — The standard deviation cannot be calculated because only one participant has been analyzed in this treatment arm at this time point.
  Week 16, n=1, 1, 2, 6, 3, 0 | 33.30 (NA) — The standard deviation cannot be calculated because only one participant has been analyzed in this treatment arm at this time point. | -14.30 (NA) — The standard deviation cannot be calculated because only one participant has been analyzed in this treatment arm at this time point. | 25.00 (35.355) | -20.08 (23.559) | -20.70 (12.804) | NA (NA) — No participants in this treatment arm were analyzed at this time point.
  Week 20, n=2, 1, 2, 6, 3, 0 | -7.65 (57.912) | -14.30 (NA) — The standard deviation cannot be calculated because only one participant has been analyzed in this treatment arm at this time point. | 9.00 (47.093) | -23.57 (27.185) | -10.97 (21.594) | NA (NA) — No participants in this treatment arm were analyzed at this time point.
  Week 24, n=1, 1, 2, 6, 3, 0 | 13.90 (NA) — The standard deviation cannot be calculated because only one participant has been analyzed in this treatment arm at this time point. | -14.30 (NA) — The standard deviation cannot be calculated because only one participant has been analyzed in this treatment arm at this time point. | 2.70 (3.818) | -19.68 (21.456) | -12.13 (21.004) | NA (NA) — No participants in this treatment arm were analyzed at this time point.

11. Secondary Outcome: Duration of Effect
Description: Duration of effect is defined as the number of days after the final injection of the FTP (after randomization in the non-treatment groups) until the date of the first recording of a value smaller than 50% in percent correction compared to the maximum change in the strabismus angle in the primary position. The strabismus angle in the primary position was measured using the APCT. The strabismus angle was evaluated as the mean value of the distant-view strabismus angle (measured at a distance of 5 m) and the near-view strabismus angle (measured at a distance of 33 cm). Percent correction compared to the maximum change in the strabismus angle was calculated as: (absolute angle [strabismus angle at Baseline minus the strabismus angle after injection]/absolute angle [strabismus angle at Baseline minus the strabismus angle at maximum change]) multiplied by 100.
Time Frame: Up to Week 48 after the final injection of the FTP (up to Study Week 52)
Population: FAS1 Population
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | BSA >=10 PD and <20 PD: Non-treatment, Then GSK1358820 | BSA >=10 PD and <20 PD: GSK1358820 1.25 U | BSA >=10 PD and <20 PD: GSK1358820 2.5 U | BSA >=20 PD and <50 PD: Non-treatment, Then GSK1358820 | BSA >=20 PD and <50 PD: GSK1358820 2.5 U | BSA >=20 PD and <50 PD: GSK1358820 5.0 U
Number analyzed (Participants) | 3 | 4 | 3 | 10 | 10 | 11
Days | 113.0 [28.0 to 231.0] | 138.0 [85.0 to NA] — The upper level of this confidence interval was not calculated because the data was censored. | 27.0 [6.0 to 63.0] | 113.5 [49.0 to 147.0] | 80.0 [25.0 to 190.0] | 84.0 [28.0 to 224.0]

12. Secondary Outcome: Severity of Duction Limitation at Weeks 1 and 4 of the FTP
Description: The severity of duction limitation was calculated for participants with paralytic strabismus. For each evaluable participant, assessment was done by taking a frontal photo of the condition of the affected eye to determine the maximum movement toward the direction to which duction is limited while the non-affected eye was masked with eye-patch. The evaluation was performed in the same eye (left or right) throughout the study period. Based on the photos, the severity of the duction limitation was assessed on a 6-point scale, with scores ranging from 0=no duction limitation to -5=cannot rotate eye to midline.
Time Frame: Week 1 and Week 4 of the FTP
Population: FAS1 Population. Only those participants available at the specified time points were analyzed (represented by n=X, X, X, X, X, X in the category titles). Different participants may have been analyzed at different time points, so the overall number of participants analyzed reflects everyone in the FAS1 Population.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Groups:
- BSA >=10 PD and <20 PD: Non-treatment: Participants (Par) with a Baseline strabismus angle (BSA) >=10 prism dioptre (PD) and <20 PD received no treatment at the start of the First Treatment Period (FTP). Par who met the additional injection criteria at 4 weeks after the start of the FTP received the injection of GSK1358820, either 1.25 Units (U) or 2.5 U, at one site of the medial rectus muscle or the lateral rectus muscle of the affected eye, then were observed for 12-24 weeks. Par who met the re-injection criteria at 12-24 weeks after the last injection (of the FTP) entered the Second Treatment Period (STP) to receive the re-injection at an appropriate dose level selected by the investigator from the prior dose level, then were observed for 24 weeks. Par who did not meet the re-injection criteria were observed for 24 more weeks. Par received a maximum of 2 injections.
- BSA >=20 PD and <50 PD: Non-treatment: Par with a BSA >=20 PD and <50 PD received no treatment at the start of the FTP. Par who met the additional injection criteria at 4 weeks after the start of the FTP received the injection of GSK1358820, either 2.5 U or 5.0 U, at one site of the medial rectus muscle or the lateral rectus muscle of the affected eye, then were observed for 12-24 weeks. Par who met the re-injection criteria at 12-24 weeks after the last injection (of the FTP) entered the STP to receive the re-injection at an appropriate dose level selected by the investigator from the prior dose level, then were observed for 24 weeks. Par who did not meet the re-injection criteria were observed for 24 more weeks. Par received a maximum of 2 injections.
Arm/Group | BSA >=10 PD and <20 PD: Non-treatment | BSA >=10 PD and <20 PD: GSK1358820 1.25 U | BSA >=10 PD and <20 PD: GSK1358820 2.5 U | BSA >=20 PD and <50 PD: Non-treatment | BSA >=20 PD and <50 PD: GSK1358820 2.5 U | BSA >=20 PD and <50 PD: GSK1358820 5.0 U
Number analyzed (Participants) | 3 | 4 | 3 | 10 | 10 | 11
Scores on a scale
  Week 1, n=0, 1, 0, 0, 1, 4 | NA (NA) — No participants in this treatment arm were analyzed at this time point. | 0.0 (NA) — The standard deviation cannot be calculated because only one participant was analyzed in this treatment arm at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point. | -1.0 (NA) — The standard deviation cannot be calculated because only one participant was analyzed in this treatment arm at this time point. | -1.3 (0.96)
  Week 4, n=0, 1, 0, 0, 1, 4 | NA (NA) — No participants in this treatment arm were analyzed at this time point. | 0.0 (NA) — The standard deviation cannot be calculated because only one participant was analyzed in this treatment arm at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point. | -1.0 (NA) — The standard deviation cannot be calculated because only one participant was analyzed in this treatment arm at this time point. | -1.0 (1.41)

13. Secondary Outcome: Severity of Duction Limitation at Weeks 1, 4, 8, 12, 16, 20, and 24 After the Final Injection of the FTP
Description: as for outcome 12
Time Frame: Weeks 1, 4, 8, 12, 16, 20, and 24 after the final injection of the FTP (up to a maximum of 52 weeks of the FTP)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | BSA >=10 PD and <20 PD: Non-treatment, Then GSK1358820 | BSA >=10 PD and <20 PD: GSK1358820 1.25 U | BSA >=10 PD and <20 PD: GSK1358820 2.5 U | BSA >=20 PD and <50 PD: Non-treatment, Then GSK1358820 | BSA >=20 PD and <50 PD: GSK1358820 2.5 U | BSA >=20 PD and <50 PD: GSK1358820 5.0 U
Number analyzed (Participants) | 3 | 4 | 3 | 10 | 10 | 11
Scores on a scale
  Week 1, n=0, 1, 0, 0, 1, 4 | NA (NA) — No participants in this treatment arm were analyzed at this time point. | 0.0 (NA) — The standard deviation cannot be calculated because only one participant was analyzed in this treatment arm at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point. | -1.0 (NA) — The standard deviation cannot be calculated because only one participant was analyzed in this treatment arm at this time point. | -1.0 (1.15)
  Week 4, n=0, 1, 0, 0, 1, 4 | NA (NA) — No participants in this treatment arm were analyzed at this time point. | 0.0 (NA) — The standard deviation cannot be calculated because only one participant was analyzed in this treatment arm at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point. | -1.0 (NA) — The standard deviation cannot be calculated because only one participant was analyzed in this treatment arm at this time point. | -1.0 (1.41)
  Week 8, n=0, 1, 0, 0, 1, 3 | NA (NA) — No participants in this treatment arm were analyzed at this time point. | 0.0 (NA) — The standard deviation cannot be calculated because only one participant was analyzed in this treatment arm at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point. | -1.0 (NA) — The standard deviation cannot be calculated because only one participant was analyzed in this treatment arm at this time point. | -1.0 (1.73)
  Week 12, n=0, 1, 0, 0, 1, 3 | NA (NA) — No participants in this treatment arm were analyzed at this time point. | 0.0 (NA) — The standard deviation cannot be calculated because only one participant was analyzed in this treatment arm at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point. | -1.0 (NA) — The standard deviation cannot be calculated because only one participant was analyzed in this treatment arm at this time point. | -0.3 (0.58)
  Week 16, n=0, 1, 0, 0, 1, 3 | NA (NA) — No participants in this treatment arm were analyzed at this time point. | 0.0 (NA) — The standard deviation cannot be calculated because only one participant was analyzed in this treatment arm at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point. | -1.0 (NA) — The standard deviation cannot be calculated because only one participant was analyzed in this treatment arm at this time point. | -0.3 (0.58)
  Week 20, n=0, 1, 0, 0, 1, 3 | NA (NA) — No participants in this treatment arm were analyzed at this time point. | 0.0 (NA) — The standard deviation cannot be calculated because only one participant was analyzed in this treatment arm at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point. | -1.0 (NA) — The standard deviation cannot be calculated because only one participant was analyzed in this treatment arm at this time point. | -0.7 (1.15)
  Week 24, n=0, 1, 0, 0, 1, 3 | NA (NA) — No participants in this treatment arm were analyzed at this time point. | 0.0 (NA) — The standard deviation cannot be calculated because only one participant was analyzed in this treatment arm at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point. | -1.0 (NA) — The standard deviation cannot be calculated because only one participant was analyzed in this treatment arm at this time point. | -0.3 (0.58)
  Week 28, n=0, 1, 0, 0, 1, 3 | NA (NA) — No participants in this treatment arm were analyzed at this time point. | 0.0 (NA) — The standard deviation cannot be calculated because only one participant was analyzed in this treatment arm at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point. | -1.0 (NA) — The standard deviation cannot be calculated because only one participant was analyzed in this treatment arm at this time point. | -0.7 (1.15)
  Week 32, n=0, 1, 0, 0, 1, 3 | NA (NA) — No participants in this treatment arm were analyzed at this time point. | 0.0 (NA) — The standard deviation cannot be calculated because only one participant was analyzed in this treatment arm at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point. | -1.0 (NA) — The standard deviation cannot be calculated because only one participant was analyzed in this treatment arm at this time point. | -0.7 (1.15)
  Week 36, n=0, 1, 0, 0, 1, 3 | NA (NA) — No participants in this treatment arm were analyzed at this time point. | 0.0 (NA) — The standard deviation cannot be calculated because only one participant was analyzed in this treatment arm at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point. | -1.0 (NA) — The standard deviation cannot be calculated because only one participant was analyzed in this treatment arm at this time point. | -0.7 (1.15)
  Week 40, n=0, 0, 0, 0, 1, 3 | NA (NA) — No participants in this treatment arm were analyzed at this time point. | NA (NA) — The standard deviation cannot be calculated because only one participant was analyzed in this treatment arm at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point. | -1.0 (NA) — The standard deviation cannot be calculated because only one participant was analyzed in this treatment arm at this time point. | -0.7 (1.15)
  Week 44, n=0, 1, 0, 0, 1, 3 | NA (NA) — No participants in this treatment arm were analyzed at this time point. | 0.0 (NA) — The standard deviation cannot be calculated because only one participant was analyzed in this treatment arm at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point. | -1.0 (NA) — The standard deviation cannot be calculated because only one participant was analyzed in this treatment arm at this time point. | -0.3 (0.58)
  Week 48, n=0, 1, 0, 0, 1, 3 | NA (NA) — No participants in this treatment arm were analyzed at this time point. | 0.0 (NA) — The standard deviation cannot be calculated because only one participant was analyzed in this treatment arm at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point. | -1.0 (NA) — The standard deviation cannot be calculated because only one participant was analyzed in this treatment arm at this time point. | -0.3 (0.58)

14. Secondary Outcome: Severity of Duction Limitation at Weeks 1, 4, 8, 12, 16, 20, and 24 of the STP
Description: The severity of duction limitation was calculated for participants with paralytic strabismus. For each evaluable participant, assessment was done by taking a frontal photo of the condition of the affected eye to determine the maximum movement toward the direction to which duction was limited while the non-affected eye was masked with eye-patch. The evaluation was performed in the same eye (left or right) throughout the study period. Based on the photos, the severity of the duction limitation was assessed on a 6-point scale, with scores ranging from 0=no duction limitation to -5=cannot rotate eye to midline. All participants with paralytic strabismus did not receive a second injection so there were no participants to analyse for this outcome measure.
Time Frame: Weeks 1, 4, 8, 12, 16, 20, and 24 of the STP (up to Study Week 52)
Population: FAS2 Population
Arm/Group | BSA >=10 PD and <20 PD: Non-treatment, Then GSK1358820 | BSA >=10 PD and <20 PD: GSK1358820 1.25 U | BSA >=10 PD and <20 PD: GSK1358820 2.5 U | BSA >=20 PD and <50 PD: Non-treatment, Then GSK1358820 | BSA >=20 PD and <50 PD: GSK1358820 2.5 U | BSA >=20 PD and <50 PD: GSK1358820 5.0 U
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

15. Secondary Outcome: Change From Baseline in the Severity of Duction Limitation at Weeks 1 and 4 of the FTP
Description: The severity of duction limitation was calculated for participants with paralytic strabismus. For each evaluable participant, assessment was done by taking a frontal photo of the condition of the affected eye to determine the maximum movement toward the direction to which duction was limited while the non-affected eye was masked with eye-patch. The evaluation was performed in the same eye (left or right) throughout the study period. Based on the photos, the severity of the duction limitation was assessed on a 6-point scale, with scores ranging from 0=no duction limitation to -5=cannot rotate eye to midline. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline and Weeks 1 and 4 of the FTP
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | BSA >=10 PD and <20 PD: Non-treatment, Then GSK1358820 | BSA >=10 PD and <20 PD: GSK1358820 1.25 U | BSA >=10 PD and <20 PD: GSK1358820 2.5 U | BSA >=20 PD and <50 PD: Non-treatment, Then GSK1358820 | BSA >=20 PD and <50 PD: GSK1358820 2.5 U | BSA >=20 PD and <50 PD: GSK1358820 5.0 U
Number analyzed (Participants) | 3 | 4 | 3 | 10 | 10 | 11
Scores on a scale
  Week 1, n=0, 1, 0, 0, 1, 4 | NA (NA) — No participants in this treatment arm were analyzed at this time point. | 0.0 (NA) — The standard deviation cannot be calculated because only one participant has been analyzed in this treatment arm at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point. | 0.0 (NA) — The standard deviation cannot be calculated because only one participant has been analyzed in this treatment arm at this time point. | 0.8 (1.71)
  Week 4, n=0, 1, 0, 0, 1, 4 | NA (NA) — No participants in this treatment arm were analyzed at this time point. | 0.0 (NA) — The standard deviation cannot be calculated because only one participant has been analyzed in this treatment arm at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point. | 0.0 (NA) — The standard deviation cannot be calculated because only one participant was analyzed in this treatment arm at this time point. | 1.0 (2.83)

16. Secondary Outcome: Change From Baseline in the Severity of Duction Limitation at Weeks 1, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, and 48 After the Final Injection of the FTP
Description: as for outcome 15
Time Frame: Baseline and Weeks 1, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, and 48 after the final injection of the FTP (up to a maximum of 52 weeks of the FTP)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | BSA >=10 PD and <20 PD: Non-treatment, Then GSK1358820 | BSA >=10 PD and <20 PD: GSK1358820 1.25 U | BSA >=10 PD and <20 PD: GSK1358820 2.5 U | BSA >=20 PD and <50 PD: Non-treatment, Then GSK1358820 | BSA >=20 PD and <50 PD: GSK1358820 2.5 U | BSA >=20 PD and <50 PD: GSK1358820 5.0 U
Number analyzed (Participants) | 3 | 4 | 3 | 10 | 10 | 11
Scores on a scale
  Week 1, n=0, 1, 0, 0, 1, 4 | NA (NA) — No participants in this treatment arm were analyzed at this time point. | 0.0 (NA) — The standard deviation cannot be calculated because only one participant has been analyzed in this treatment arm at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point. | 0.0 (NA) — The standard deviation cannot be calculated because only one participant was analyzed in this treatment arm at this time point. | 1.0 (1.41)
  Week 4, n=0, 1, 0, 0, 1, 4 | NA (NA) — No participants in this treatment arm were analyzed at this time point. | 0.0 (NA) — The standard deviation cannot be calculated because only one participant has been analyzed in this treatment arm at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point. | 0.0 (NA) — The standard deviation cannot be calculated because only one participant was analyzed in this treatment arm at this time point. | 1.0 (2.83)
  Week 8, n=0, 1, 0, 0, 1, 3 | NA (NA) — No participants in this treatment arm were analyzed at this time point. | 0.0 (NA) — The standard deviation cannot be calculated because only one participant has been analyzed in this treatment arm at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point. | 0.0 (NA) — The standard deviation cannot be calculated because only one participant was analyzed in this treatment arm at this time point. | 1.7 (3.06)
  Week 12, n=0, 1, 0, 0, 1, 3 | NA (NA) — No participants in this treatment arm were analyzed at this time point. | 0.0 (NA) — The standard deviation cannot be calculated because only one participant has been analyzed in this treatment arm at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point. | 0.0 (NA) — The standard deviation cannot be calculated because only one participant was analyzed in this treatment arm at this time point. | 2.3 (2.31)
  Week 16, n=0, 1, 0, 0, 1, 3 | NA (NA) — No participants in this treatment arm were analyzed at this time point. | 0.0 (NA) — The standard deviation cannot be calculated because only one participant has been analyzed in this treatment arm at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point. | 0.0 (NA) — The standard deviation cannot be calculated because only one participant was analyzed in this treatment arm at this time point. | 2.3 (2.31)
  Week 20, n=0, 1, 0, 0, 1, 3 | NA (NA) — No participants in this treatment arm were analyzed at this time point. | 0.0 (NA) — The standard deviation cannot be calculated because only one participant has been analyzed in this treatment arm at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point. | 0.0 (NA) — The standard deviation cannot be calculated because only one participant was analyzed in this treatment arm at this time point. | 2.0 (2.65)
  Week 24, n=0, 1, 0, 0, 1, 3 | NA (NA) — No participants in this treatment arm were analyzed at this time point. | 0.0 (NA) — The standard deviation cannot be calculated because only one participant has been analyzed in this treatment arm at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point. | 0.0 (NA) — The standard deviation cannot be calculated because only one participant was analyzed in this treatment arm at this time point. | 2.3 (2.31)
  Week 28, n=0, 1, 0, 0, 1, 3 | NA (NA) — No participants in this treatment arm were analyzed at this time point. | 0.0 (NA) — The standard deviation cannot be calculated because only one participant has been analyzed in this treatment arm at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point. | 0.0 (NA) — The standard deviation cannot be calculated because only one participant was analyzed in this treatment arm at this time point. | 2.0 (2.65)
  Week 32, n=0, 1, 0, 0, 1, 3 | NA (NA) — No participants in this treatment arm were analyzed at this time point. | 0.0 (NA) — The standard deviation cannot be calculated because only one participant has been analyzed in this treatment arm at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point. | 0.0 (NA) — The standard deviation cannot be calculated because only one participant was analyzed in this treatment arm at this time point. | 2.0 (2.65)
  Week 36, n=0, 1, 0, 0, 1, 3 | NA (NA) — No participants in this treatment arm were analyzed at this time point. | 0.0 (NA) — The standard deviation cannot be calculated because only one participant has been analyzed in this treatment arm at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point. | 0.0 (NA) — The standard deviation cannot be calculated because only one participant was analyzed in this treatment arm at this time point. | 2.0 (2.65)
  Week 40, n=0, 0, 0, 0, 1, 3 | NA (NA) — No participants in this treatment arm were analyzed at this time point. | NA (NA) — The standard deviation cannot be calculated because only one participant has been analyzed in this treatment arm at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point. | 0.0 (NA) — The standard deviation cannot be calculated because only one participant was analyzed in this treatment arm at this time point. | 2.0 (2.65)
  Week 44, n=0, 1, 0, 0, 1, 3 | NA (NA) — No participants in this treatment arm were analyzed at this time point. | 0.0 (NA) — The standard deviation cannot be calculated because only one participant has been analyzed in this treatment arm at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point. | 0.0 (NA) — The standard deviation cannot be calculated because only one participant was analyzed in this treatment arm at this time point. | 2.3 (2.31)
  Week 48, n=0, 1, 0, 0, 1, 3 | NA (NA) — No participants in this treatment arm were analyzed at this time point. | 0.0 (NA) — The standard deviation cannot be calculated because only one participant has been analyzed in this treatment arm at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point. | 0.0 (NA) — The standard deviation cannot be calculated because only one participant was analyzed in this treatment arm at this time point. | 2.3 (2.31)

17. Secondary Outcome: Change From Baseline in the Severity of Duction Limitation at Weeks 1, 4, 8, 12, 16, 20, and 24 of the STP
Description: The severity of duction limitation was calculated for participants with paralytic strabismus. For each evaluable participant, assessment was done by taking a frontal photo of the condition of the affected eye to determine the maximum movement toward the direction to which duction was limited while the non-affected eye was masked with eye-patch. The evaluation was performed in the same eye (left or right) throughout the study period. Based on the photos, the severity of the duction limitation was assessed on a 6-point scale, with scores ranging from 0=no duction limitation to -5=cannot rotate eye to midline. Change from Baseline was calculated as the post-Baseline value minus the Baseline value. All participants with paralytic strabismus did not receive a second injection so there were no participants to analyse for this outcome measure.
Time Frame: Baseline and Weeks 1, 4, 8, 12, 16, 20, and 24 of the STP (up to Study Week 52)
Population: FAS2 Population
Arm/Group | BSA >=10 PD and <20 PD: Non-treatment, Then GSK1358820 | BSA >=10 PD and <20 PD: GSK1358820 1.25 U | BSA >=10 PD and <20 PD: GSK1358820 2.5 U | BSA >=20 PD and <50 PD: Non-treatment, Then GSK1358820 | BSA >=20 PD and <50 PD: GSK1358820 2.5 U | BSA >=20 PD and <50 PD: GSK1358820 5.0 U
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious adverse events (AEs) reported from the start of randomization up to Week 24 of the FTP are summarized.
Description: SAEs and non-serious AEs were summarized for members of the Safety Population (SP1), comprised of all randomized participants in the FTP.
Groups:
- Non-treatment: Participants (par) with a BSA of greater than or equal to 10 PD and less than 20 PD or greater than or equal to 20 PD and less than 50 PD received no treatment from the start of the First Treatment Period (FTP). Par were re-evaluated at Week 4 and Weeks 12-24. Par who did not meet the injection criteria at any time point remained in the FTP group and were observed up to study Week 52.
- Non-treatment, Then GSK1358820: Par with a BSA of greater than or equal to 10 PD and less than 20 PD or greater than or equal to 20 PD and less than 50 PD received no treatment from the start of the FTP. Par who met the additional injection criteria at 4 weeks after the start of the FTP received the injection of GSK1358820, either 1.25 Units (U), 2.5 U, or 5.0 U at one site of the medial rectus muscle or the lateral rectus muscle of the affected eye, then were observed for 12-24 weeks. Par who met the re-injection criteria at 12-24 weeks after the last injection (of the FTP) entered the Second Treatment Period (STP) to receive the re-injection at an appropriate dose level selected by the investigator from the prior dose level, then were observed for 24 weeks. Par who did not meet the re-injection criteria were observed for 24 more weeks. Par received a maximum of 2 injections.
- GSK1358820 1.25 U: Par with a BSA greater than or equal to 10 PD and less than 20 PD received the first injection of GSK1358820 1.25 U at one site of the medial rectus muscle or the lateral rectus muscle of the affected eye at the start of the FTP. Par who met the additional injection criteria at 4 weeks after the start of the FTP received an additional injection of GSK1358820, either 1.25 U or 2.5 U, at the same site and in the same eye as the previous injection, then were observed for 12-24 weeks. Par who met the re-injection criteria at 12-24 weeks after the last injection (of the FTP) entered the STP to receive the re-injection at an appropriate dose level selected by the investigator from the prior dose level, then were observed for 24 weeks. Par who did not meet the re-injection criteria were observed for 24 more weeks. Par received a maximum of 3 injections.
- GSK1358820 2.5 U: Participants with BSA of greater than or equal to 10 PD and less than 20 PD or greater than or equal to 20 PD and less than 50 PD received the first injection of GSK1358820 2.5 U at one site of the medial rectus muscle or the lateral rectus muscle of the affected eye at the start of the FTP. Par who met the additional injection criteria at 4 weeks after the start of the FTP received an additional injection of GSK1358820, either 2.5 U or 5.0, at the same site and in the same eye as the previous injection, then were observed for 12-24 weeks. Par who met the re-injection criteria at 12-24 weeks after the last injection (of the FTP) entered the STP to receive the re-injection at an appropriate dose level selected by the investigator from the prior dose level, then were observed for 24 weeks. Par who did not meet the re-injection criteria were observed for 24 more weeks. Par received a maximum of 3 injections.
- GSK1358820 5.0 U: Par with a BSA greater than or equal to 20 PD and less than 50 PD received the first injection of GSK1358820 5.0 U at one site of the medial rectus muscle or the lateral rectus muscle of the affected eye at the start of the FTP. Par who met the additional injection criteria at 4 weeks after the start of the FTP received an additional injection of GSK1358820, either 5.0 U or 10.0 U, at the same site and in the same eye as the previous injection, then were observed for 12-24 weeks. Par who met the re-injection criteria at 12-24 weeks after the last injection (of the FTP) entered the STP to receive the re-injection at an appropriate dose level selected by the investigator from the prior dose level, then were observed for 24 weeks. Par who did not meet the re-injection criteria were observed for 24 more weeks. Par received a maximum of 3 injections.
Arm/Group | Non-treatment | Non-treatment, Then GSK1358820 | GSK1358820 1.25 U | GSK1358820 2.5 U | GSK1358820 5.0 U
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13 | 0/4 | 1/13 | 0/11
Other Adverse Events (participants affected / at risk) | 1/13 | 8/13 | 1/4 | 6/13 | 6/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Non-treatment (N=13) | Non-treatment, Then GSK1358820 (N=13) | GSK1358820 1.25 U (N=4) | GSK1358820 2.5 U (N=13) | GSK1358820 5.0 U (N=11)
Strabismus (Eye disorders) | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Non-treatment (N=13) | Non-treatment, Then GSK1358820 (N=13) | GSK1358820 1.25 U (N=4) | GSK1358820 2.5 U (N=13) | GSK1358820 5.0 U (N=11)
Eyelid ptosis (Eye disorders) | 0 | 3 | 0 | 2 | 2
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 0 | 1 | 1
Conjunctival hyperaemia (Eye disorders) | 0 | 0 | 0 | 2 | 0
Diplopia (Eye disorders) | 0 | 1 | 0 | 0 | 1
Eye movement disorder (Eye disorders) | 0 | 1 | 0 | 0 | 0
Strabismus (Eye disorders) | 0 | 0 | 0 | 0 | 1
Conjunctival deposit (Eye disorders) | 0 | 0 | 0 | 1 | 0
Conjunctivitis allergic (Eye disorders) | 0 | 0 | 1 | 0 | 0
Corneal erosion (Eye disorders) | 0 | 1 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 1 | 0
Ophthalmoplegia (Eye disorders) | 0 | 1 | 0 | 0 | 0
Punctate keratitis (Eye disorders) | 0 | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 1 | 0 | 2 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 2 | 0 | 0 | 0
Helicobacter infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Dental caries (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Therapeutic response increased (General disorders) | 0 | 0 | 0 | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Periorbital contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Liver function test abnormal (Investigations) | 0 | 0 | 0 | 1 | 0
Calculus urinary (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Vertigo positional (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.